CLINICAL TRIAL: NCT03810664
Title: A Phase 1, Single-Center, Randomized, Cross-Over, Clinical Study Investigating the Comparability of Somatrogon in Two Different Drug Product Presentations
Brief Title: A Clinical Study Investigating the Comparability of Somatrogon in Two Different Drug Product Presentations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CP-4-011
Record Dates: First submitted 2019-01-08; First posted 2019-01-22 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — somatrogon

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, single-center, open-label randomized, 2×2 crossover (Ref Test | Test Ref) study with a washout of two weeks to establish bioequivalence between single dose of somatrogon in a PEN to somatrogon in VIAL administered sc in healthy male volunteers.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Somatrogon pre-filled PEN (Experimental)
  Interventions: Drug: Somatrogon
- Somatrogon frozen liquid formulation (Active Comparator)
  Interventions: Drug: Somatrogon

INTERVENTIONS:
Drug: Somatrogon — A single dose of 12 mg of somatrogon will be injected as one sc injection to the arm on each dosing day (Day 0 and Day 14).

SUMMARY:
This is a Phase 1, single-center, open-label randomized, 2×2 crossover (Ref Test | Test Ref) study with a washout of two weeks to establish bioequivalence between single dose of somatrogon in a PEN to somatrogon in VIAL administered sc in healthy male volunteers.

DETAILED DESCRIPTION:
The subjects will undergo a screening period (Day -28 to -1), and when eligible for study participation will be randomized to receive one sc injection of one of two somatrogon drug product presentations on Day 0, either the PEN or VIAL presentation. A series of blood draws and study procedures will be carried out over the course of the next 10 days to evaluate the subjects. Following a two week washout period, the subjects will be brought back to the clinic to receive the other somatrogon drug product presentation, and once again followed for the next 14 days to study completion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-55 (inclusive) years
* Body Mass Index (BMI) 19 to 32 kg/m2 (inclusive) and weighing at least 55 kg
* Non-smoking (by declaration) for a period of at least six months prior to screening visit

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male volunteers
Enrollment: 49 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the serum concentration-time from time 0 to a specific time (AUCt) | 30 days
Area under the curve (AUC) of the serum concentration-time from time 0 to infinity (AUC∞) | 30 days
Serum concentration from of maximum concentration (Cmax) of somatrogon levels in serum | 30 days

SECONDARY OUTCOMES:
AUCt of IGF-1 and IGFBP-3 levels | 30 days
AUC∞ of IGF-1 and IGFBP-3 levels | 30 days
Cmax of IGF-1 and IGFBP-3 levels | 30 days
Time to maximum concentration (Tmax) | 30 days
Apparent Terminal Rate Constant (λz) and t½ | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Pagnusset, MD, Principal Investigator — QPS Miami Research Associates
Locations (1):
- QPS Miami Research Associates, Miami, Florida, United States